CLINICAL TRIAL: NCT06314113
Title: Evaluation of Oral Epigallocatechin Gallate Treatment for Low-grade Cervical Lesions (L-SIL) Associated With Human Papilloma Virus (HPV) Infection
Brief Title: Evaluation of Oral EGCG Treatment for L-SIL Associated With HPV Infection
Acronym: EGCG-HPV
Status: Recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Palermo
Other Study IDs: EGCG-HPV
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Low-Grade Intraepithelial Neoplasia of Cervix
Keywords: Human Papilloma Virus (HPV); Low-Grade Intraepithelial Neoplasia of Cervix; Epigallocatechin Gallate
MeSH Terms: interventions — epigallocatechin gallate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low-grade Cervical Lesions (L-SIL): Women affected by Low-grade Cervical Lesions (L-SIL) associated with Human Papilloma Virus (HPV) Infection
  Interventions: Dietary Supplement: Epigallocatechin Gallate

INTERVENTIONS:
Dietary Supplement: Epigallocatechin Gallate — Oral treatment with Epigallocatechin Gallate 200 mg per day

SUMMARY:
The study aims to evaluate the effectiveness of the synergy of oral Epigallocatechin Gallate as a treatment for Low-grade Cervical Lesions (L-SIL) associated with Human Papilloma Virus (HPV) infection.

DETAILED DESCRIPTION:
Human papilloma virus (HPV) infection is the most widespread infection worldwide among the sexually active population. Papillomaviruses are a very large and heterogeneous family of double-stranded DNA viruses (8kb). They have no envelope and have icosahedral symmetry. Their viral genome is divided into two regions defined as 1) early and 2) late. The early genes encode the early proteins E1, E2, E4, E5, E6, E7 necessary for viral DNA replication and cellular transformation. The late genes encode the late proteins L1, L2 which serve for the formation of the viral capsid. HPV viruses are classified based on their oncogenicity. Those at low risk are associated with proliferative lesions, generally benign, of the skin and mucous membranes. The clinical manifestations include common, flat and plantar warts, genital and flat condylomata acuminata which are the result of sexual transmission of the virus and which arise on the penis, anus, female genitalia, urethra, perianal area and straight. High-risk HPVs, on the other hand, are those that integrate into the host's genome and cause lesions that can evolve into carcinoma over time. However, it has recently been shown that even viruses normally defined as low risk can cause precancerous lesions in the case of tumors of the vulva, vagina, penis and anus. In 80% of cases the infection resolves spontaneously within two years, however in 20% of cases, the infection persists and causes the onset of lesions of varying degrees which over time can evolve into neck cancer of the uterus in women or penile cancer in men. In fact, if HPV is now recognized as the etiological agent of cervical cancer in 99.7% of cases, it is estimated that it is also responsible for 50% of penile tumors and 26-30% of cord tumors oral.

Persistence therefore represents an oncological risk factor for those who contract the infection, since if the infection persists for over a year, there is a high probability that the viral DNA integrates into the host's genome. Integration involves the constitutive expression of some viral oncoproteins (E6/E7) that block the activity of host tumor suppressor genes (p53/pRB). The blockade of tumor suppressors in turn stimulates an uncontrolled proliferation of lesions, which, due to a failure to activate the inhibitory regulatory processes of our organism, leads to tumor development.

In the case of lesions classified as "low grade" (L-SIL), the common practice is to check the patient after six months, while in the case of lesions classified as "high grade" (H-SIL), the therapeutic standard is represented by the surgical removal of these lesions. However, removal of the lesion does not guarantee total eradication of the infection, as the virus could persist in the adjacent healthy mucosa. Currently, there are no treatments against HPV infection, nor against the persistence of the virus. Various types of therapies are associated with primary (vaccination) and secondary (screening programs) prevention programs for the treatment of clinical manifestations induced by the virus, such as warts. Among the treatments that are used as normal clinical practice in the field of HPV infections, also for the treatment of warts, those based on epigallocatechin gallate (EGCG) represent a novelty that has been proven to be safe and effective.

Epigallocatechin gallate (EGCG), the main polyphenolic component of green tea, has antioxidant, anti-inflammatory and anticancer properties. Its action has also been extensively tested on cervical cancer lines, on which EGCG exerts an antiproliferative and pro-apoptotic action in a dose-dependent manner. A recent study demonstrated that EGCG increases the expression levels of p53 protein and reduces the levels of viral oncoproteins E6/E7. A randomized clinical trial has also highlighted how treatment with EGCG has a chemo-preventive action on the progression of lesions in HPV-positive women with lesions of various degrees, leading to a reduction in the degree of the lesions themselves.

Considering these elements, the study aims to evaluate the effectiveness of the synergy of oral Epigallocatechin Gallate as a treatment for Low-grade Cervical Lesions (L-SIL) associated with Human Papilloma Virus (HPV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by Low-grade Cervical Lesions (L-SIL) associated with Human Papilloma Virus (HPV) Infection

Exclusion Criteria:

* Pregnancy
* Concomitant pathologies causing immunosuppression
* Concurrent Immunomodulatory therapies
* Hormone replacement therapy
* High-grade Cervical Lesions (H-SIL) or in situ adenocarcinoma
* Previous history of L-SIL or higher grade lesions ≥ 24 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women affected by Low-grade Cervical Lesions (L-SIL) associated with Human Papilloma Virus (HPV) Infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Persistence | After 6, 12, 18, and 24 months from the recruitment
  Persistence of Low-grade Cervical Lesions (L-SIL), evaluated by pap smear

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — University of Palermo; Giuseppe Mascellino, M.D., Study Chair — University of Palermo; Pietro Serra, M.D., Study Chair — University of Palermo; Andrea Etrusco, M.D., Study Chair — University of Palermo
Locations (1):
- "Paolo Giaccone" Hospital, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No